CLINICAL TRIAL: NCT00148902
Title: A Phase I, Open-Label Study of the Safety, Tolerability and Pharmacokinetics of GW572016 in Combination With Docetaxel (Taxotere)
Brief Title: Effects Of GW572016 In Combination With Docetaxel (TAXOTERE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGF10021
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Neoplasms, Breast
Keywords: tumor
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Lapatinib; Docetaxel

ARMS (1):
- All treated subjects (Experimental): All subjects received Lapatinib in Combination with Docetaxel (Taxotere)
  Interventions: Drug: lapatinib; Drug: docetaxel

INTERVENTIONS:
Drug: lapatinib — lapatinib
Drug: docetaxel — docetaxel

SUMMARY:
This is a safety and tolerability study of GW572016 given with docetaxel (TAXOTERE).

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumors.
* Able to swallow oral medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-04-28 (Actual); Primary Completion 2006-01-21 (Actual); Study Completion 2006-01-21 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs) or serious AEs (SAEs) | Up to 7 weeks in each cycle
  An AE is any untoward medical occurrence in a subject or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require medical or surgical intervention will be categorized as SAE.
Number of subjects with abnormal change from Baseline in laboratory parameters | Baseline and up to 7 weeks in each cycle
  Blood sample will be collected to evaluate laboratory parameters.
Number of subjects with Optimally Tolerated regimen | Up to 7 weeks in each cycle
  Optimally Tolerated regimen is a dose regimen where 1 out of 6 subjects experiences a dose-limiting toxicity (DLT).

SECONDARY OUTCOMES:
Area under the plasma drug concentration curve (AUC) from 0 to infinity (AUC[0-inf]) of docetaxel alone (Pharmacokinetic [PK] cohort 1) | Sequence 1, Day 1 and Sequence 2, Day 22: Prior to the docetaxel infusion, at 20 and 40 minutes after the start of the infusion, at 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours after start of the infusion.
  Blood samples will be collected at indicated time points to evaluate pharmacokinetic parameters.
AUC within the dosing interval (AUC[0-tau]) of GW572016 alone (PK cohort 2) | Sequence 1, Day 1 and Sequence 2, Day 21: Prior to GW572016 dose and at 20 and 40 minutes; 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours after the dose.
  Blood samples will be collected at indicated time points to evaluate pharmacokinetic parameters.
AUC (0-tau) of GW572016 when given in combination with docetaxel (PK cohort 1) | Sequence 1, Day 22 and Sequence 2, Day 1: Prior to the GW572016 oral dose and docetaxel infusion, at 20 and 40 minutes after the start of the infusion, at 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours after the start of the docetaxel infusion.
  Blood samples will be collected at indicated time points to evaluate pharmacokinetic parameters.
AUC (0-tau) of GW572016 when given in combination with docetaxel (PK cohort 2) | Sequence 1, Day 23 and Sequence 2, Day 1: Prior to the GW572016 oral dose and docetaxel infusion, at 20 and 40 minutes after the start of the infusion, at 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours after the start of the docetaxel infusion
  Blood samples will be collected at indicated time points to evaluate pharmacokinetic parameters.
Maximum observed plasma drug concentration (Cmax) of docetaxel alone (PK cohort 1) | Sequence 1, Day 1 and Sequence 2, Day 22: Prior to the docetaxel infusion, at 20 and 40 minutes after the start of the infusion, at 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours after start of the infusion.
  Blood samples will be collected at indicated time points to evaluate pharmacokinetic parameters.
Cmax of GW572016 alone (PK cohort 2) | Sequence 1, Day 1 and Sequence 2, Day 21: Prior to GW572016 dose and at 20 and 40 minutes; 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours after the dose.
  Blood samples will be collected at indicated time points to evaluate pharmacokinetic parameters.
Cmax of GW572016 when given in combination with docetaxel (PK cohort 1) | Sequence 1, Day 22 and Sequence 2, Day 1: Prior to the GW572016 oral dose and docetaxel infusion, at 20 and 40 minutes after the start of the infusion, at 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours after the start of the docetaxel infusion.
  Blood samples will be collected at indicated time points to evaluate pharmacokinetic parameters.
Cmax of GW572016 when given in combination with docetaxel (PK cohort 2) | Sequence 1, Day 23 and Sequence 2, Day 1: Prior to the GW572016 oral dose and docetaxel infusion, at 20 and 40 minutes after the start of the infusion, at 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours after the start of the docetaxel infusion
  Blood samples will be collected at indicated time points to evaluate pharmacokinetic parameters.
Time to maximum observed plasma drug concentration (Tmax) of docetaxel alone (PK cohort 1) | Sequence 1, Day 1 and Sequence 2, Day 22: Prior to the docetaxel infusion, at 20 and 40 minutes after the start of the infusion, at 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours after start of the infusion.
  Blood samples will be collected at indicated time points to evaluate pharmacokinetic parameters.
Tmax of GW572016 alone (PK cohort 2) | Sequence 1, Day 1 and Sequence 2, Day 21: Prior to GW572016 dose and at 20 and 40 minutes; 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours after the dose.
  Blood samples will be collected at indicated time points to evaluate pharmacokinetic parameters.
Tmax of GW572016 when given in combination with docetaxel (PK cohort 1) | Sequence 1, Day 22 and Sequence 2, Day 1: Prior to the GW572016 oral dose and docetaxel infusion, at 20 and 40 minutes after the start of the infusion, at 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours after the start of the docetaxel infusion.
  Blood samples will be collected at indicated time points to evaluate pharmacokinetic parameters.
Tmax of GW572016 when given in combination with docetaxel (PK cohort 2) | Sequence 1, Day 23 and Sequence 2, Day 1: Prior to the GW572016 oral dose and docetaxel infusion, at 20 and 40 minutes after the start of the infusion, at 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours after the start of the docetaxel infusion
  Blood samples will be collected at indicated time points to evaluate pharmacokinetic parameters.
Concentration at the last measurable time point (Ctau) for GW572016 along (PK cohort 2) | Sequence 1, Day 1 and Sequence 2, Day 21: Prior to GW572016 dose and at 20 and 40 minutes; 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours after the dose.
  Blood samples will be collected at indicated time points to evaluate pharmacokinetic parameters.
Time to first measurable plasma drug concentration (Tlag) for GW572016 along (PK cohort 2) | Sequence 1, Day 1 and Sequence 2, Day 21: Prior to GW572016 dose and at 20 and 40 minutes; 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours after the dose.
  Blood samples will be collected at indicated time points to evaluate pharmacokinetic parameters.
AUC from time zero to time of last measurable concentration (AUClast) for docetaxel alone (PK cohort 1) | Sequence 1, Day 1 and Sequence 2, Day 22: Prior to the docetaxel infusion, at 20 and 40 minutes after the start of the infusion, at 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours after start of the infusion.
  Blood samples will be collected at indicated time points to evaluate pharmacokinetic parameters.
Clearance (CL) for docetaxel alone (PK cohort 1) | Sequence 1, Day 1 and Sequence 2, Day 22: Prior to the docetaxel infusion, at 20 and 40 minutes after the start of the infusion, at 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours after start of the infusion.
  Blood samples will be collected at indicated time points to evaluate pharmacokinetic parameters.
Volume of distribution at steady state (Vss) for docetaxel alone (PK cohort 1) | Sequence 1, Day 1 and Sequence 2, Day 22: Prior to the docetaxel infusion, at 20 and 40 minutes after the start of the infusion, at 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours after start of the infusion.
  Blood samples will be collected at indicated time points to evaluate pharmacokinetic parameters.
Elimination half-life (Thalf) for docetaxel alone (PK cohort 1) | Sequence 1, Day 1 and Sequence 2, Day 22: Prior to the docetaxel infusion, at 20 and 40 minutes after the start of the infusion, at 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours after start of the infusion.
  Blood samples will be collected at indicated time points to evaluate pharmacokinetic parameters.
Number of subjects with complete response | Week 3 of every third cycle
  Efficacy assessments will be obtained every three cycles depending on standard practices in specific tumor type.
Number of subjects with partial response | Week 3 of every third cycle
  Efficacy assessments will be obtained every three cycles depending on standard practices in specific tumor type.
Number of subjects with stable disease | Week 3 of every third cycle
  Efficacy assessments will be obtained every three cycles depending on standard practices in specific tumor type.
Number of subjects with progressive disease | Week 3 of every third cycle
  Efficacy assessments will be obtained every three cycles depending on standard practices in specific tumor type.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Nashville, Tennessee

REFERENCES:
- See also: Results for study EGF10021 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/EGF10021?search=study&study_ids=EGF10021#rs